CLINICAL TRIAL: NCT02257385
Title: Study DB2116961, A Multicentre, Randomised, Blinded, Parallel Group Study to Compare UMEC/VI (Umeclidinium/Vilanterol) in a Fixed Dose Combination With Indacaterol Plus Tiotropium in Symptomatic Subjects With Moderate to Very Severe COPD
Brief Title: Comparative Study of Umeclidinium/Vilanterol (UMEC/VI) in a Fixed Dose Combination With Indacaterol Plus Tiotropium
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 116961
Record Dates: First submitted 2014-10-02; First posted 2014-10-06 (Estimated); Results first posted 2016-03-03 (Estimated); Last update posted 2018-03-01 (Actual); Status verified 2018-02

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: indacaterol; efficacy; FEV1; ELLIPTA; non inferiority; vilanterol; COPD; safety; tiotropium; umeclidinium bromide; GSK573719
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Tiotropium Bromide; indacaterol; Albuterol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- UMEC/VI arm (Experimental): Participants will be instructed to self-administer one dose each morning of UMEC/VI Inhalation Powder 62.5/25 mcg once daily via ELLIPTA DPI, placebo once daily via HANDIHALER inhaler and placebo once daily via BREEZHALER inhaler
  Interventions: Drug: UMEC/VI; Drug: UMEC/VI matching placebo; Drug: Albuterol/salbutamol Metered Dose Inhaler (MDI)
- Tiotropium + Indacaterol arm (Placebo Comparator): Participants will be instructed to self-administer one dose each morning of Tiotropium bromide 18 mcg once daily via HANDIHALER inhaler, Indacaterol 150 mcg once daily via BREEZHALER inhaler and placebo once daily via ELLIPTA DPI
  Interventions: Drug: Tiotropium; Drug: Tiotropium matching placebo; Drug: Indacaterol; Drug: Indacaterol matching placebo; Drug: Albuterol/salbutamol Metered Dose Inhaler (MDI)

INTERVENTIONS:
Drug: UMEC/VI — ELLIPTA DPI will be supplied with 30 doses (2 strips with 30 blisters per strip) where first strip contains Umeclidinium bromide (unit dose strengths 62.5 mcg per blister) blended with lactose monohydrate and magnesium stearate 0.6% weight/weight (w/w) of total drug product and second strip contains Vilanterol (unit dose strengths 25 mcg per blister) blended with lactose monohydrate and magnesium stearate 1.0% w/w of total drug product
  Arms: UMEC/VI arm
Drug: UMEC/VI matching placebo — ELLIPTA DPI will be supplied with 30 doses (2 strips with 30 blisters per strip) where first strip contains lactose monohydrate and magnesium stearate 0.6% w/w of total drug product and second strip contains lactose monohydrate and magnesium stearate 1.0% w/w of total drug product
  Arms: UMEC/VI arm
Drug: Tiotropium — Tiotropium (as bromide monohydrate) inhalation capsules 18 mcg per dose will be supplied along with HANDIHALER inhalers manufactured by Boehringer Ingelheim
  Arms: Tiotropium + Indacaterol arm
Drug: Tiotropium matching placebo — Tiotropium matching placebo capsules manufactured by GSK, will contain lactose and will be supplied along with HANDIHALER inhalers
  Arms: Tiotropium + Indacaterol arm
Drug: Indacaterol — Indacaterol inhalation capsules 150 mcg per dose will be supplied by GSK along with BREEZHALER inhalers manufactured by Novartis
  Arms: Tiotropium + Indacaterol arm
Drug: Indacaterol matching placebo — Indacaterol matching placebo capsules manufactured by GSK, will contain lactose and will be supplied along with BREEZHALER inhalers manufactured by Novartis
  Arms: Tiotropium + Indacaterol arm
Drug: Albuterol/salbutamol Metered Dose Inhaler (MDI) — Albuterol/salbutamol MDI or nebules for as needed use will be issued throughout the study. Albuterol/salbutamol will be sourced from local commercial stock. If not available locally, GSK will source centrally

SUMMARY:
This is a Phase IIIb multicentre, randomised, blinded, triple dummy, parallel group study to evaluate the efficacy and safety of UMEC/VI inhalation powder (62.5/25 microgram [mcg] Once daily [QD]) when administered via ELLIPTA® Dry Powder Inhaler (DPI) compared to indacaterol plus tiotropium (150 mcg/18 mcg respectively QD) administered via individual inhalers over a treatment period of 12 weeks in participants with moderate to very severe Chronic Obstructive Pulmonary Disease (COPD). The purpose of this study is to demonstrate that UMEC/VI (delivered via ELLIPTA DPI), when used in symptomatic moderate to very severe COPD participants, is non-inferior to the combination of indacaterol (delivered via BREEZHALER® inhaler) plus tiotropium (delivered via HANDIHALER® inhaler) on measures of trough forced expiratory volume in one second (FEV1) after 12 weeks of treatment. Participants who met the eligibility criteria at screening (Visit 1) will complete a 5 to 7 day run in period prior to randomisation at Visit 2. Clinic visits will follow at day 2, week 2, week 4, week 8 and week 12 of treatment, plus week 12 + 1 day (Visits 3 to 8). The total duration of study participation will be approximately 14 weeks. ELLIPTA is a registered trademark of the GSK group of companies. HANDIHALER is a registered trademark of Boehringer Ingelheim Pharma GmbH & Co. KG. BREEZHALER is a registered trademark of Novartis AG.

ELIGIBILITY:
Inclusion Criteria:

* Type of subject: Outpatient
* Informed Consent: A signed and dated written informed consent prior to study participation.
* Participants 40 years of age or older at Visit 1.
* Gender: Male or female participants. A female is eligible to enter and participate in the study if she is of: Non-child bearing potential (i.e., physiologically incapable of becoming pregnant, including any female who is post-menopausal or surgically sterile). Surgically sterile females are defined as those with a documented hysterectomy and/or bilateral oophorectomy or tubal ligation. Post-menopausal females are defined as being amenorrhoeic for greater than 1 year with an appropriate clinical profile, e.g., age appropriate, > 45 years, in the absence of hormone replacement therapy.OR Child bearing potential, has a negative pregnancy test at screening, and agrees to one of the following acceptable contraceptive methods used consistently and correctly (i.e., in accordance with the approved product label and the instructions of the physician for the duration of the study screening to follow-up contact): Abstinence, Oral Contraceptive, either combined or progestogen alone, Injectable progestogen, Implants of levonorgestrel, Estrogenic vaginal ring, Percutaneous contraceptive patches, Intrauterine device (IUD) or intrauterine system (IUS) that meets the Standard Operating Procedure (SOP) effectiveness criteria as stated in the product label, Male partner sterilization (vasectomy with documentation of azoospermia) prior to the female subject's entry into the study, and this male is the sole partner for that subject. For this definition, "documented" refers to the outcome of the investigator's/designee's medical examination of the subject or review of the subject's medical history for study eligibility, as obtained via a verbal interview with the subject or from the subject' s medical records. Double barrier method: condom and an occlusive cap (diaphragm or cervical/vault caps) with a vaginal spermicidal agent (foam/gel/film/cream/suppository)
* Diagnosis: An established clinical history of COPD in accordance with the definition by the American Thoracic Society/European Respiratory Society.
* Smoking History: Current or former cigarette smokers with a history of cigarette smoking of >=10 pack-years. Former smokers are defined as those who have stopped smoking for at least 6 months prior to Visit 1.
* Severity of Disease: A pre and post-albuterol/salbutamol Forced Expiratory Volume in One Second/ Forced Vital Capacity (FEV1/ FVC) ratio of <0.70 and a pre and post-albuterol/salbutamol FEV1 of <=70% predicted normal value at Visit 1, calculated using Quanjer reference equations.
* Dyspnoea: A score of >= 2 on the Modified Medical Research Council Dyspnoea Scale (mMRC) at Visit 1.
* QT interval corrected (QTc) Criteria: QTc <450 milliseconds (msec) or QTc <480 msec for patients with bundle branch block The QTc is the QT interval corrected for heart rate according to either Bazett's formula (QTcB), Fridericia's formula (QTcF), or another method, machine or manual overread. For subject eligibility and withdrawal, QTcF will be used. For purposes of data analysis, QTcF will be used as primary. The QTc should be based on single or averaged QTc values of triplicate Electrocardiogram (ECGs) obtained over a brief recording period.
* French participants: In France, a subject will be eligible for inclusion in this study only if either affiliated to or a beneficiary of a social security category.

Exclusion Criteria:

* Pregnancy: Women who are pregnant or lactating or are planning on becoming pregnant during the study.
* Asthma: A current diagnosis of asthma.
* Other Respiratory Disorders: Known alpha-1 antitrypsin deficiency, active lung infections (such as tuberculosis), and lung cancer are absolute exclusionary conditions. A subject who, in the opinion of the investigator, has any other significant respiratory conditions in addition to COPD should be excluded. Examples may include clinically significant bronchiectasis, pulmonary hypertension, sarcoidosis, or interstitial lung disease. Allergy rhinitis is not exclusionary.
* Other Diseases/Abnormalities: Participants with historical or current evidence of clinically significant cardiovascular, neurological, psychiatric, renal, hepatic, immunological, endocrine (including uncontrolled diabetes or thyroid disease) or hematological abnormalities that are uncontrolled and/or a previous history of cancer in remission for <5 years prior to Visit 1 (localized carcinoma of the skin that has been resected for cure is not exclusionary). Significant is defined as any disease that, in the opinion of the investigator, would put the safety of the subject at risk through participation, or which would affect the efficacy or safety analysis if the disease/condition exacerbated during the study.
* Contraindications: A history of allergy or hypersensitivity to any anticholinergic/muscarinic receptor antagonist, beta2-agonist, lactose/milk protein or magnesium stearate or a medical condition such as narrow-angle glaucoma, prostatic hypertrophy or bladder neck obstruction that, in the opinion of the study physician, contraindicates study participation or use of an inhaled anticholinergic or beta 2 agonist.
* Hospitalisation: Hospitalisation for COPD or pneumonia within 12 weeks prior to Visit 1.
* Lung Resection: Participants with lung volume reduction surgery within the 12 months prior to Screening (Visit 1).
* 12-Lead ECG: An abnormal and significant ECG finding from the 12-lead ECG conducted at Visit 1. Specific ECG findings that preclude subject eligibility will be listed in protocol The study investigator will determine the medical significance of any ECG abnormalities not listed.
* Screening labs: Significantly abnormal finding from clinical chemistry or haematology tests at Visit 1 as determined by the study investigator.
* Medication Prior to Spirometry: Unable to withhold albuterol/salbutamol for the 4 hour period required prior to spirometry testing at each study visit.
* Medications prior to Screening: Use of the following medications according to the following defined time intervals prior to Visit 1: Depot corticosteroids (12 weeks); Oral or parenteral corticosteroids (6 weeks); Antibiotics (for lower respiratory tract infection) (6 weeks); Cytochrome P450 3A4 strong inhibitors ( 6 weeks); Long Acting Beta-Agonist (LABA)/ inhaled corticosteroids (ICS) combination products (e.g. fluticasone/salmeterol, mometasone, furoate/formoterol fumarate, budesonide/formoterol, fumarate), If LABA/ICS therapy is discontinued completely (30 days); If discontinuing LABA therapy and switching to ICS monotherapy (48 hours for salmeterol or formoterol, 14 days for Olodaterol, Indacaterol or, Vilanterol); Use of ICS at a dose >1000 mcg/day of fluticasone propionate or equivalent (30 days); Initiation or discontinuation of ICS use (30 days); Inhaled long acting beta2-agonists (LABA): Salmeterol, Formoterol (48 hours), Olodaterol, Indacaterol and Vilanterol (14 days); Long acting muscarinic antagonists (LAMA) (Tiotropium, Aclidinium, Glycopyrronium, Umeclidinium) (7 days); LABA/LAMA combination products (Whichever mono component has the longest washout); Roflumilast (14 days); Oral beta-agonists- Long-acting (48 hours), Short-acting(12 hours); Theophyllines (48 hours); Oral leukotriene inhibitors (zafirlukast, montelukast, zileuton) (48 hours); Inhaled sodium cromoglycate or nedocromil sodium (24 hours); Inhaled short acting beta2-agonists (4 hours); Inhaled short-acting anticholinergic (short acting muscarinic antagonist [SAMA]) products eg ipratropium (4 hours); Inhaled short-acting anticholinergic/short-acting beta2-agonist combination products (SAMA/Short Acting beta2-agonists [SABA]) (4 hours); Any other investigational medication (30 days or within 5 drug half-lives)
* Oxygen: Use of Long Term Oxygen Therapy (LTOT).This is defined as oxygen therapy prescribed for greater than 12 hours per day. As needed oxygen use (i.e. <=12 hours per day) is not exclusionary.
* Nebulized Therapy: Regular use (prescribed for use every day, not for as-needed use) of short-acting bronchodilators (e.g., albuterol/salbutamol) via nebulized therapy.
* Pulmonary Rehabilitation Program: Participation in the acute phase of a pulmonary rehabilitation program within 12 weeks prior to Visit 1. Participants who are in the maintenance phase of a pulmonary rehabilitation program are not excluded.
* Drug or Alcohol Abuse: A known or suspected history of alcohol or drug abuse within 2 years prior to Visit 1.
* Affiliation with Investigator Site: Is an investigator, sub-investigator, study coordinator, employee of a participating investigator or study site, or immediate family member of the aforementioned that is involved in this study.
* Inability to read: In the opinion of the investigator, any subject who is unable to read and/or would not be able to complete a questionnaire.
* Participants who are pre-screen or screen failures cannot be re-screened.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 967 (Actual)
Dates: Start 2014-10-15 (Actual); Primary Completion 2015-05-04 (Actual); Study Completion 2015-05-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (66):
- Argentina (5):
  - GSK Investigational Site, Mar del Plata, Buenos Aires
  - GSK Investigational Site, San Miguel de Tucumán, Tucumán Province
  - GSK Investigational Site, Buenos Aires
  - GSK Investigational Site, Mendoza
  - GSK Investigational Site, San Miguel de Tucumán
- Chile (3):
  - GSK Investigational Site, Puente Alto - Santiago, Región Metro de Santiago
  - GSK Investigational Site, Santiago, Región Metro de Santiago
  - GSK Investigational Site, Santiago
- Estonia (2):
  - GSK Investigational Site, Haapsalu
  - GSK Investigational Site, Tallinn
- France (6):
  - GSK Investigational Site, Gières
  - GSK Investigational Site, Nantes
  - GSK Investigational Site, Perpignan
  - GSK Investigational Site, Reims
  - GSK Investigational Site, Strasbourg
  - GSK Investigational Site, Tarbes
- Germany (6):
  - GSK Investigational Site, Rüdersdorf, Brandenburg
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Schwerin, Mecklenburg-Vorpommern
  - GSK Investigational Site, Magdeburg, Saxony-Anhalt
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Hamburg
- Hungary (8):
  - GSK Investigational Site, Balassagyarmat
  - GSK Investigational Site, Budaörs
  - GSK Investigational Site, Debrecen
  - GSK Investigational Site, Gödöllő
  - GSK Investigational Site, Nyíregyháza
  - GSK Investigational Site, Pécs
  - GSK Investigational Site, Szeged
  - GSK Investigational Site, Szikszó
- Italy (5):
  - GSK Investigational Site, Piacenza, Emilia-Romagna
  - GSK Investigational Site, Pordenone, Friuli Venezia Giulia
  - GSK Investigational Site, Mantova, Lombardy
  - GSK Investigational Site, Tradate (VA), Lombardy
  - GSK Investigational Site, Novara, Piedmont
- Peru (2):
  - GSK Investigational Site, Lima, Lima Province
  - GSK Investigational Site, Lima
- Poland (6):
  - GSK Investigational Site, Elblag
  - GSK Investigational Site, Krakow
  - GSK Investigational Site, Ostrów Wielkopolski
  - GSK Investigational Site, Piekary Śląskie
  - GSK Investigational Site, Sopot
  - GSK Investigational Site, Słupsk
- Romania (5):
  - GSK Investigational Site, Bucharest
  - GSK Investigational Site, Cluj-Napoca
  - GSK Investigational Site, Constanța
  - GSK Investigational Site, Râmnicu Vâlcea
  - GSK Investigational Site, Timișoara
- Russia (13):
  - GSK Investigational Site, Arkhangelsk
  - GSK Investigational Site, Irkutsk
  - GSK Investigational Site, Kazan'
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Omsk
  - GSK Investigational Site, Orenburg
  - GSK Investigational Site, Perm
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Saint Petesburg
  - GSK Investigational Site, Stavropol
  - GSK Investigational Site, Tomsk
  - GSK Investigational Site, Ulyanovsk
  - GSK Investigational Site, Yekaterinburg
- Slovakia (5):
  - GSK Investigational Site, Bojnice
  - GSK Investigational Site, Humenné
  - GSK Investigational Site, Poprad
  - GSK Investigational Site, Spišská Nová Ves
  - GSK Investigational Site, Vráble

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Kalberg C, O'Dell D, Galkin D, Newlands A, Fahy WA. Dual Bronchodilator Therapy with Umeclidinium/Vilanterol Versus Tiotropium plus Indacaterol in Chronic Obstructive Pulmonary Disease: A Randomized Controlled Trial. Drugs R D. 2016 Jun;16(2):217-27. doi: 10.1007/s40268-016-0131-2. PMID 27028749
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: 116961 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 116961 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 116961 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 116961 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 116961 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 116961 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 116961 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible participants (par) completed a 5-7 day run-in period, and were randomized to blinded study medication for 12 weeks. Supplemental albuterol/salbutamol was provided to all par, to be used on an as-needed basis during run-in and up to Day 85.
Pre-assignment Details: A total of 1190 par were screened; 967 par randomized and 961 par comprised the Intent-to-Treat (ITT) Population (Pop), comprised of all par randomized to treatment (trt) who received at least 1 dose of randomized study medication in the trt period.
Groups:
- Umeclidinium/Vilanterol 62.5/25 µg: Participants self-administered one dose each morning from each of the following three inhalers for 12 weeks: ELLIPTA dry powder inhaler containing umeclidinium/vilanterol inhalation powder 62.5/25 micrograms (µg), BREEZHALER containing placebo, and HANDIHALER containing placebo. Each inhaler containing placebo was identical in appearance to its corresponding inhaler containing active study medication.
- Indacaterol 150 µg + Tiotropium Bromide 18 µg: Participants self-administered one dose each morning from each of the following three inhalers for 12 weeks: ELLIPTA dry powder inhaler containing placebo, BREEZHALER containing indacaterol 150 µg, and HANDIHALER containing tiotropium bromide 18 µg. The inhaler containing placebo was identical in appearance to its corresponding inhaler containing active study medication.
Period: Overall Study
Arm/Group | Umeclidinium/Vilanterol 62.5/25 µg | Indacaterol 150 µg + Tiotropium Bromide 18 µg
Started | 482 | 479
Completed | 460 | 457
Not Completed | 22 | 22
Not completed — Adverse Event | 12 | 8
Not completed — Lack of Efficacy | 1 | 2
Not completed — Protocol Violation | 5 | 7
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Umeclidinium/Vilanterol 62.5/25 µg | Indacaterol 150 µg + Tiotropium Bromide 18 µg | Total
Number analyzed (Participants) | 482 | 479 | 961
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.4 (7.75) | 64.0 (8.44) | 64.2 (8.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 127 | 138 | 265
  Male | 355 | 341 | 696
Race/Ethnicity, Customized [Number; unit: Participants]
  American Indian or Alaska Native | 24 | 27 | 51
  Asian - Central/South Asian Heritage | 1 | 0 | 1
  Asian - East Asian Heritage | 0 | 1 | 1
  Asian - Japanese Heritage | 4 | 1 | 5
  White - Arabic/North African Heritage | 0 | 1 | 1
  White -White/Caucasian/European Heritage | 453 | 449 | 902

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Trough Forced Expiratory Volume in One Second (FEV1) on Treatment Day 85 (Visit 8)
Description: FEV1 is a measure of lung function and is defined as the maximal amount of air that can be forcefully exhaled in 1 second. BL was the mean of the 2 assessments made 30 and 5 minutes (min) pre-dose (PD) on Day 1. Trough FEV1 measurements were taken electronically by spirometry on Days 2, 28, 56, 84 and 85. Trough FEV1 on Day 85 is defined as the mean of the FEV1 values obtained at 23 and 24 hours (hr) after dosing on Day 84 (at Week 12 + 1 day). Analysis was performed using mixed model repeated measures (RM) with covariates of trt, BL FEV1 (mean of values measured at 30 and 5 min PD on Day 1), center group, day, day by BL interaction and day by trt interaction, where day was nominal.
Time Frame: Baseline (BL) and Day 85
Population: Per Protocol (PP) Pop: all ITT Pop par who were not full protocol deviators considered to impact efficacy. Only par with data available at the specified time points (TP) were analyzed but all par without (w/o) missing covariate information and with >= 1 post BL measurement were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Umeclidinium/Vilanterol 62.5/25 µg | Indacaterol 150 µg + Tiotropium Bromide 18 µg
Number analyzed (Participants) | 392 | 392
Liters | 0.172 (0.0107) | 0.171 (0.0108)
Statistical Analysis 1: Comparison: Umeclidinium/Vilanterol 62.5/25 µg vs Indacaterol 150 µg + Tiotropium Bromide 18 µg; Test type: Non-Inferiority or Equivalence — Alternate hypothesis:the difference between the trt means (umeclidinium/vilanterol minus indacaterol + tiotropium bromide) would be > -50 milliliters (mL). If the lower CI (2.5% 1-sided significance level) of the statistical test should fall above -50 mL, then umeclidinium/vilanterol may be deemed statistically non-inferior to indacaterol plus tiotropium. If the lower CI (2.5% 1-sided significance) of the statistical testing exceeded 0 then, statistical superiority would have been established; p = 0.964, Mixed Models Analysis; Least Squares Mean Difference = 0.001, 95% CI 2-sided [-0.029 to 0.030]

2. Secondary Outcome: Change From Baseline in Weighted Mean (WM) FEV1 Over 0-6 Hour Post-dose at Day 84
Description: BL FEV1 was the mean of the 2 assessments made 30 and 5 min PD on Day 1. WM FEV1 derived by calculating the area under the FEV1/time curve (AUC) using the trapezoidal rule, and then dividing the value by the time interval over which the AUC was calculated. The WM was calculated at Days 1 and 84 using the 0-6 hr post-dose FEV1 measurements collected on that day, which included PD FEV1 (taken 30 and 5 min prior to dosing on Day 1 and the 30 and 5 min reading prior to dosing on Day 84) and post-dose FEV1 measurements at 1, 3 and 6 hr post-dose.WM change from BL was the WM at at the visit minus the BL value. Analysis was performed using a RM model with covariates of trt, BL FEV1 (mean of values measured at 30 and 5 min PD on Day 1) center group, day, day by BL and day by trt interaction, where day was nominal. Only par with data available at the specified TP were analyzed but all par w/o missing covariate information and with >=1 post-BL measurement were included in the analysis.
Time Frame: Baseline and Day 84
Population: ITT Population
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Umeclidinium/Vilanterol 62.5/25 µg | Indacaterol 150 µg + Tiotropium Bromide 18 µg
Number analyzed (Participants) | 455 | 452
Liters | 0.235 (0.0111) | 0.258 (0.0111)
Statistical Analysis 1: Comparison: Umeclidinium/Vilanterol 62.5/25 µg vs Indacaterol 150 µg + Tiotropium Bromide 18 µg; Test type: Superiority or Other; p = 0.145, Mixed Models Analysis; Least Squares Mean Difference = -0.023, 95% CI 2-sided [-0.054 to 0.008]

ADVERSE EVENTS:
Time Frame: On-treatment serious adverse events (SAEs) and non-serious adverse events (AEs) were collected over a period of a maximum of 96 days starting from Day 1 of treatment until the follow-up contact.
Description: On-treatment SAEs and non-serious AEs were reported for members of the ITT Population, comprised of all participants randomized to treatment who received at least one dose of randomized study medication in the treatment period.
Arm/Group | Umeclidinium/Vilanterol 62.5/25 µg | Indacaterol 150 µg + Tiotropium Bromide 18 µg
Serious Adverse Events (participants affected / at risk) | 21/482 | 16/479
Other Adverse Events (participants affected / at risk) | 76/482 | 65/479
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Umeclidinium/Vilanterol 62.5/25 µg (N=482) | Indacaterol 150 µg + Tiotropium Bromide 18 µg (N=479)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 6 | 3
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia (Infections and infestations) | 2 | 2
Gastroenteritis (Infections and infestations) | 1 | 0
Laryngitis (Infections and infestations) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Angina pectoris (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
Atrioventricular block (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 0 | 1
Ventricular fibrillation (Cardiac disorders) | 1 | 0
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma of the oral cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Epilepsy (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Circulatory collapse (Vascular disorders) | 1 | 0
Peripheral artery thrombosis (Vascular disorders) | 0 | 1
Peripheral ischaemia (Vascular disorders) | 1 | 0
Crohn's disease (Gastrointestinal disorders) | 1 | 0
Chest pain (General disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Umeclidinium/Vilanterol 62.5/25 µg (N=482) | Indacaterol 150 µg + Tiotropium Bromide 18 µg (N=479)
Headache (Nervous system disorders) | 36 (56) | 28 (60)
Nasopharyngitis (Infections and infestations) | 32 (34) | 27 (31)
Cough (Respiratory, thoracic and mediastinal disorders) | 16 (18) | 17 (18)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.